CLINICAL TRIAL: NCT05170438
Title: Phase II Trial of Lenvatinib Plus Paclitaxel for Patients With Advanced Biliary Tract Cancer Who Failed to Gemcitabine-based Treatment
Brief Title: Lenvatinib Plus Paclitaxel for Patients With Advanced Biliary Tract Cancer Who Failed to Gemcitabine-based Treatment
Acronym: LenPac
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); China Medical University, Taiwan (Other); Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1222
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Cancer
Keywords: Biliary Tract Cancer; Gemcitabine; Lenvatinib
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: 1.Safety run-in phase: 3-6 cases Traditional 3+3 design is applied for the determination of initial lenvatinib dose.2 Extension phase:3.
  The estimated number of patients in current trial is calculated with Simon's minimax two-stage analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib 12 or 16 mg/day orally,D28; Paclitaxel 80 mg/m2 in 250-500 mL of NS, IV D 1, 8, 15; (Experimental): one arm Lenvatinib 16 or 12 mg/day orally day 1-28; Paclitaxel 80 mg/m2 in 250-500 mL of normal saline, intravenously over 2 hours on day 1, 8, 15;
  Interventions: Drug: Lenvatinib Pill,Paclitaxel

INTERVENTIONS:
Drug: Lenvatinib Pill,Paclitaxel — Regimen Every 28 days as one cycle.Lenvatinib 16 or 12 mg/day orally (depends on the result of safety run-in phase), on day 1-28; Paclitaxel 80 mg/m2 in 250-500 mL of normal saline, intravenously over 2 hours on day 1, 8, 15.

SUMMARY:
To evaluate the following items in patients with advanced cholangiocarcinoma receiving lenvatinib plus paclitaxel treatment, Primary endpoint: Overall response rate (ORR) by RECIST 1.1 Secondary endpoints Progression-free survival (PFS) Time to progression Overall survival Disease control rate (Overall response rate + stable disease ≧ 4 weeks) Response rate by modified RECIST Association between therapeutic efficacy and tumor vascularity Quality of life Safety profile Predictive biomarker of cholangiocarcinoma

DETAILED DESCRIPTION:
1. Safety run-in phase: 2-6 cases Traditional 3+3 design is applied for the determination of initial lenvatinib dose.
2. Extension phase:

   The estimated number of patients in current trial is calculated with Simon's minimax two-stage analysis. Considering the response rate is at least 10% higher (based on Ueno's data) than the 5% response rate of mFOLFOX in patients who fail gemcitabine plus cisplatin in ABC-06 trial, the assumption of response rate of lenvatinib plus paclitaxel will is 15% or higher. Therefore, Simon's minimax two-stage design is applied with P0 = 5%, P1 = 15%, error 0.10, and errors 0.20. If tumor response is not observed in the first 29 patients, the study will be stopped. Otherwise, 15 additional patients be accrued for a total of 44. The null hypothesis will be rejected if 5 or more subjects have tumor response to the treatment of lenvatinib plus paclitaxel in 44 patients. If the investigators assume that drop-out rate is 10%, total accrual patient will be 49.
3. Total case number = patients in safety run-in phase + patients in extension phase = (2 - 6) + 49 = 51 - 55

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with age ≧20 years old.
* 2.Histologically confirmed biliary tract cancer which is locally advanced, recurrent or metastatic disease. The disease entities include intrahepatic cholangiocarcinoma, perihilar cholangiocarcinoma, distal bile duct cholangiocarcinoma, Ampulla of Vater cancer, and gallbladder cancer.

  3.Documented disease progression during or within 6 months after gemcitabine-based (regimens containing gemcitabine plus cisplatin, gemcitabine plus S-1, or gemcitabine plus oxaliplatin) chemotherapy. Patient who has received antiangiogenetic agent (bevacizumab, ramucirumab, lenvatinib), taxane-based chemotherapy, or more than 1 line of chemotherapy for locally advanced or metastatic biliary tract cancer is ineligible.

  4. Documented measurable disease as defined by RECIST v1.1. 5. Baseline Eastern Cooperative Oncology Group performance status score 0-1. 6. Patient has life expectancy of at least 12 weeks. 7. Adequate hematologic parameters, and hepatic and renal functions defined as 7.1: Hepatic: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 2.5 x upper limit of normal (ULN) ( 5.0 x ULN if attributable to liver metastases), total bilirubin 3 mg/dL.

7.2: Renal: serum creatinine level 1.5 x ULN or creatinine clearance > 30 ml/min [calculated by either Cockcroft-Gault equation [(140-age) x body weight (kg) x (1 if male or 0.85 if female) / (72 x serum creatinine level, mg/dl)] or 24-hour urine test].

7.3: Hematological: white blood cell 3,000/ul, absolute neutrophil count (ANC) 1,500/ul, hemoglobin 9 g/dl and platelet count 90,000/ul.

8. Adequate controlled blood pressure (BP), defined as BP≦140/90 mmHg at screening and no change in antihypertensive medication within 1 week prior to the cycle1/day 1.

9. Adequate blood coagulation function, defined as prothrombin time international normalized ratio (PT INR)≦ 2.3.

10. Normal ECG or ECG without any clinical significant findings 11. Able to understand and sign an informed consent (or have a legal representative who is able to do so).

12. Women or men of reproductive potential should agree to use an effective contraceptive method

Exclusion Criteria:

* 1. Patients who have major abdominal surgery, radiotherapy or other investigating agents within 2 weeks are not eligible. Patients who have palliative radiotherapy will be eligible if the irradiated area does not involve the only lesion of measurable / evaluable disease.

  2. Patients having liver dysfunction with Child-Pugh score ≧7. 3. Patients with gastrointestinal malabsorption or condition that might affect the absorption of lenvatinib in the opinion of the investigator.

  4. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. Patients with tumor invasion/infiltration of major blood vessels should be excluded because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following therapy.

  5. Uncontrolled blood pressure (systolic BP>140 mmHg or diastolic BP>90 mmHg) in spite of an optimized regimen of antihypertensive medication.

  6. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months, or cardiac arrhythmia requiring medical treatment.

  7. Patients having > 1+ proteinuria on urine dipstick testing will undergo 24 h urine collection for quantitative assessment of proteinuria. Subjects with urine protein≧ 1 g/24 h will be ineligible.

  8. Patients with electrolyte abnormalities that have not been corrected. 9. Patients with metastatic lesion in central nervous system. 10. Patients with active infection. 11. Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy.

  12. Patients who have peripheral neuropathy > grade I of any etiology 13. Patients who have serious concomitant systemic disorders incompatible with the study, i.e. poorly controlled diabetes mellitus, auto-immune disorders, or other condition that in the opinion of the investigator would preclude the subject's participation in the study.

  14. Patients who have other prior or concurrent malignancy except for adequately treated in situ carcinoma or basal cell carcinoma of skin, or any malignancy which remains disease-free for 3 or more years after curative treatment.

  15. Females who are breastfeeding or pregnant at screening or baseline. 16. Patients with psychiatric illness which would preclude study compliance.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 year
  Overall response rate (ORR) by RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 year
  Progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Yuan Bai, MD,PhD, Study Chair — China Medical University Hospital; Tsang-Wu Liu, MD, Study Director — Taiwan Cooperative Oncology Group, National Health Research Institutes
Locations (8):
- Taiwan (8):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No